CLINICAL TRIAL: NCT01854060
Title: Predictive Factors for a Clinical Diagnosis of Irritable Bowel Syndrome in a Large Cohort of 440,822 Young Adults.
Brief Title: Predictive Factors for a Clinical Diagnosis of Irritable Bowel Syndrome in a Large Cohort of Young Adults.
Status: Completed | Type: Observational
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, DAN CARTER, Head of Gastro Service, Medical Corps, Israel Defense Force
Other Study IDs: IDF-1083-2011
Record Dates: First submitted 2013-05-12; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Epidimiology; Deterioration in the severity of irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- irritable bowel syndrome: All new cases of clinical diagnosis of irritable bowel syndrome

SUMMARY:
The prevalence of IBS in the community has been reported in numerous cross-sectional surveys. However, less is known about the incidence of IBS ,mainly due to its slow development and to patients under-reporting. Furthermore, only one study has analyzed data concerning potential risk factors for the diagnosis of IBS. The investigators will examine the incidence of IBS in a large cohort of young adults and will look at the association of socioeconomic, anthropometric and occupational factors with IBS incidence.

ELIGIBILITY:
Inclusion Criteria:

* All Israeli men and women
* aged 18-39 years
* served in active military service (mandatory and career service) between the years 2005-2011

Exclusion Criteria:

* Diagnosis of celiac disease
* Inflammatory bowel disease
* Cancer in the digestive system

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of Israeli men and women aged 18-39 years who served in active military service (mandatory and career service) between the years 2005-2011
Sampling Method: Non-Probability Sample
Enrollment: 440822 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical diagnosis of irritable bowel syndrome | 6 years
  New diagnosis of irritable bowel syndrome during this priod

SECONDARY OUTCOMES:
predictive factors for the clinical diagnosis of irritable bowel syndrome | 6 years
  Anthropometric and demographic factors predictive for the clinicaldiagnosis of irritable bowel syndrome including gender, body mass index, ethnicity , type of service

CONTACTS AND LOCATIONS:
Locations (1):
- Israel Defence Forces, Medical Corps, Ramat Gan, Israel